CLINICAL TRIAL: NCT03978507
Title: Digital Wearable Walking Aid for Freezing of Gait in Parkinson´s Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: KU Leuven (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-18-NG-0908-18-TLV-CTIL
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease
Keywords: Freezing of Gait; Intelligent external cueing systems; Free living gait monitoring; Patient-Adaptive Freezing of Gait Detection System
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is an interventional study with a parallel design, consisting of pre- and post-assessments, 2x (pre- and post) 7 days of free-living gait monitoring and an intervention/control period of 4 weeks. The pre-assessment and first week of free-living gait monitoring will take place prior to randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Prior to randomization, all participants will be informed that the goal of the study is to compare the effects of two types of feedback about physical activity on freezing of gait. By withholding information about the cueing intervention, we hope that the participants in the control group will not realize that they are in the control group, in order to avoid a lack of motivation in this group. The intervention group will probably become unmasked after group allocation, as the cueing therapy was not mentioned in the informed consent.
  During the post-assessment, the FOG provoking protocol will be performed with and without cueing. This induces the risk of the investigator/outcome assessor becoming unmasked, as patients in the control group may mention that this cueing option is something they haven't experienced during the intervention period. In order to prevent this, the therapist will ask patients in the intervention group to also act surprised to the cueing modality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DeFOG group (Experimental): feedback number of steps + cueing
  Interventions: Behavioral: Intelligent cueing; Behavioral: Feedback about the number of steps
- Control group (Active Comparator): feedback number of steps
  Interventions: Behavioral: Feedback about the number of steps

INTERVENTIONS:
Behavioral: Intelligent cueing — 1 month use of an intelligent, wearable device that provides personalized cueing only when FOG is detected
  Arms: DeFOG group
Behavioral: Feedback about the number of steps — Feedback about the number of steps is given in the intervention group as well as in the control group during the 1-month intervention-period.

SUMMARY:
The objective of this study is to investigate the effects of relatively long-term use of a wearable device that provides personalized and intelligent cues (e.g. only when FOG is detected) on FOG.

DETAILED DESCRIPTION:
The objective of this study is to investigate the effects of relatively long-term use of a wearable device that provides personalized and intelligent cues (e.g. only when FOG is detected) on FOG. It is hypothesized that the use of this device will reduce FOG in the home and in the community more than in a group of freezers who only receive basic gait information unrelated to FOG-episodes.

This study is a single- blinded bi-centric randomized controlled trial, consisting of 4 weeks of intervention, pre- and post- assessments and free-living monitoring. For this purpose, the DeFOG system was developed through a collaboration between our research group, the Sourasky Medical Center Tel Aviv and mHealth Technologies Bologna, Italy. The system consists of a smartphone, 2 foot-mounted inertial measurement units (IMU's) and earphones which enable transmitting feedback and auditory cues for gait, when FOG is about to occur. The patients will be randomized into an intervention group (DeFOG group) or a control group (N=31 per group). All patients will wear the DeFOG system (mHealth Technologies, mHT) and both groups will receive feedback about the daily number of steps produced. But, only the DeFOG group will receive cueing following detection of FOG. The cueing consists of a metronome, and if FOG persists, also a verbal instruction will be delivered. A therapist will personalize the settings of the DeFOG system and will support the patients in using the system (for instance in coping with false positives). Pre- and post- assessments will be performed by a blinded researcher, both before and after taking medication (in OFF and ON medication state, respectively), consisting of FOG-provoking tasks and questionnaires. During the post-assessment, the FOG provoking protocol will be repeated in both groups with and without the cueing option of the DeFOG system in the home situation.

If therapists involved in the trial note an increase of falls throughout the trial, then it can be decided to involve an interim analysis of the data monitoring committee.

ELIGIBILITY:
Inclusion criteria:

1. Clinical diagnosis of Parkinson's disease (PD) (n=31 per site) according to the UK PD Society Brain Bank criteria
2. Modified Hoehn & Yahr Stage I to IV in the ON-state;
3. Age between 40 and 90 years;
4. Ability to walk 5 minutes while unassisted by another person;
5. Mini-Mental State Examination (MMSE) score of >= 21 or > 16 on the 26-item MMSE screening;
6. Stable PD medication during the previous month and no medication change foreseen for the next 6 weeks.
7. Self-reported freezing of gait (FOG) severity of at least 1 FOG episode per day, based on Characterizing of Freezing of Gait Questionnaire, irrespective of FOG occurring ON- or OFF-medication.

Exclusion criteria:

1. Participation in another clinical study;
2. Use of a cueing device as normal practice;
3. A fall frequency of more than once a day;
4. Acute musculoskeletal or other neurological or cardiovascular conditions affecting gait or any other medical condition which, in the opinion of the investigator, may prevent completing the protocol;
5. Hearing problems, precluding use of auditory feedback from the DeFOG system;
6. The occurrence of any of the following within 3 months prior to informed consent: orthopedic surgery of the lower extremity, myocardial infarction, hospitalization for unstable angina, coronary artery bypass graft, percutaneous coronary intervention, implantation of a cardiac resynchronization therapy device, implantation of deep brain stimulation;
7. Substance abuse, major depressive disorder or clinical apathy that affects daily walking activity or may interfere with the patient's compliance;
8. Inability to walk without a rollator indoors;
9. Use of a Duodopa® or apomorphine injections, jeopardizing OFF-medication assessments;
10. Absence of clinically observed FOG during the FOG-provoking assessment at the pre-intervention assessment (T1).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in severity of the freezing of gait phenomenon: percentage time frozen (%TF) | immediate post-intervention
  %TF is determined based on video annotations of the full FOG-provoking protocol (OFF+ON) during the pre- and post-intervention assessment (T1 and T2). %TF = (summed duration FOG during FOG-provoking protocol ON+OFF)/(total duration FOG-provoking protocol OFF+ON)*100%. Freezing includes episodes of akinetic FOG, trembling FOG and festination.

SECONDARY OUTCOMES:
Changes in severity of the freezing of gait phenomenon: %TF OFF medication | immediate post-intervention
  %TF is determined based on video annotations of the OFF-phase of the FOG-provoking protocol during the pre- and post-intervention assessment (T1 and T2). %TF = (summed duration FOG during FOG-provoking protocol OFF)/(total duration FOG-provoking protocol OFF)*100%. Freezing includes episodes of akinetic FOG, trembling FOG and festination.
Changes in severity of the freezing of gait phenomenon: %TF ON medication | immediate post-intervention
  %TF is determined based on video annotations of the ON-phase of the FOG-provoking protocol during the pre- and post-intervention assessment (T1 and T2). %TF = (summed duration FOG during FOG-provoking protocol ON)/(total duration FOG-provoking protocol ON)*100%. Freezing includes episodes of akinetic FOG, trembling FOG and festination.
Change in number and duration of FOG episodes (video-based) | immediate post-intervention
  The number and duration of FOG episodes as determined based on annotations of video recordings of the FOG-provoking protocol, both OFF and ON medication, during the pre- and post-intervention assessment (T1 and T2).
Changes in severity of the freezing of gait phenomenon (subjective measurement): score on new Freezing of Gait questionnaire (NFOG-Q). | immediate post-intervention
  The change in the score on the New Freezing of Gait questionnaire (NFOG-Q), which is the revised version of the original Freezing of Gait Questionnaire. The NFOG-Q consists of 9 items, and the maximum score is 28. Higher scores correspond to more severe perceived FOG. The NFOG-Q is administered during the pre- and post-intervention assessments (T1 and T2).
Changes in physical activity, as recorded using an accelerometer placed on the lower back. | One week post-intervention
  Physical activity will be determined based on recordings using an accelerometer placed on the lower back for 7 days (Axivity; AX3: 3-Axis Logging Accelerometer or AX6: 6-Axis Logging Accelerometer). Outcome measures include the number of steps, the number of bouts of physical activity and the duration of bouts of physical activity. The Axivity sensor is placed before the start of the pre- and post intervention assessment (T1 and T2) and will record continuously for 7 days (during the monitoring weeks).
Changes in Timed Up and Go (TUG) test Performance (sec) | immediate post-intervention
  Change in the duration to perform the Timed-Up and Go (TUG) test in seconds, with and without a cognitive dual task (serial-3 subtraction), both OFF- and ON-medication. The Timed Up and Go performance is a measure of mobility, and a longer duration to perform the task represents a more impaired mobility. The TUG test is administered as part of the FOG-provoking protocol, during the pre- and post-intervention assessments (T1 and T2).
Changes in 4 meter walk test (4MW) performance (sec) | immediate post-intervention
  Change in the duration to walk 4 meters (in seconds), both OFF- and ON-medication. The full 4 meter walk test (4MW) back and forth with turn consists of 5 meters (0.5 meter acceleration, 4 meter steady state walking, 0.5 meter deceleration, a turn on the spot, and then again 0.5 meter acceleration, 4 meter steady state walking and 0.5 meter deceleration). The duration to walk 4 meters before and after the turn will be determined based on video annotations and averaged. The 4MW is administered as part of the FOG-provoking protocol, during the pre- and post-intervention assessments (T1 and T2).
Change in motor function: score on the MDS-UPDRS part III | immediate post-intervention
  Score on the Motor Examination (part III) of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), assessed both OFF and ON-medication during the pre- and post-intervention assessments (T1 and T2). MDS-UPDRS is a tool to measure the severity and progression of Parkinson disease (PD). Part III is a motor examination consisting of 14 items, each rated on a 5-point Likert type scale (ranging from 0 to 4), with higher scores indicating more severe impairment. The maximum UPDRS part III score is 132, with higher score representing worse motor disability from PD.
Change in balance: score on the MiniBESTest | immediate post-intervention
  Change in score on the Mini-Balance Evaluation Systems Test (MiniBESTest), as assessed during the pre- and post-intervention assessment while ON-medication. The MiniBESTest consists of 14 items designed to measure balance performance during mobility tasks related to daily activities. Each item receives a score of 0 to 2, where a score of 0 represents an inability to complete the item and a score of 2 represents the ability to complete the task independently. The range of scores is 0-28, with a higher score representing worse balance impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Hausdorff, PhD, Study Chair — Tel-Aviv Sourasky Medical Center
Locations (2):
- Catholic University (KU) Leuven, Leuven, Flamish-Brabant, Belgium
- Labrotory for Gait and Neurodynamics, Movement Disorders Unit, TASMC, Tel Aviv, IL, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Palmerini L, Rocchi L, Mazilu S, Gazit E, Hausdorff JM, Chiari L. Identification of Characteristic Motor Patterns Preceding Freezing of Gait in Parkinson's Disease Using Wearable Sensors. Front Neurol. 2017 Aug 14;8:394. doi: 10.3389/fneur.2017.00394. eCollection 2017. PMID 28855887
- [Background] Mazilu S, Calatroni A, Gazit E, Mirelman A, Hausdorff JM, Troster G. Prediction of Freezing of Gait in Parkinson's From Physiological Wearables: An Exploratory Study. IEEE J Biomed Health Inform. 2015 Nov;19(6):1843-54. doi: 10.1109/JBHI.2015.2465134. Epub 2015 Aug 5. PMID 26259206
- [Background] Ginis P, Nieuwboer A, Dorfman M, Ferrari A, Gazit E, Canning CG, Rocchi L, Chiari L, Hausdorff JM, Mirelman A. Feasibility and effects of home-based smartphone-delivered automated feedback training for gait in people with Parkinson's disease: A pilot randomized controlled trial. Parkinsonism Relat Disord. 2016 Jan;22:28-34. doi: 10.1016/j.parkreldis.2015.11.004. PMID 26777408
- [Background] Sweeney D, Quinlan LR, Browne P, Richardson M, Meskell P, OLaighin G. A Technological Review of Wearable Cueing Devices Addressing Freezing of Gait in Parkinson's Disease. Sensors (Basel). 2019 Mar 13;19(6):1277. doi: 10.3390/s19061277. PMID 30871253
- [Background] Mancini M, Bloem BR, Horak FB, Lewis SJG, Nieuwboer A, Nonnekes J. Clinical and methodological challenges for assessing freezing of gait: Future perspectives. Mov Disord. 2019 Jun;34(6):783-790. doi: 10.1002/mds.27709. Epub 2019 May 2. PMID 31046191
- [Derived] Denk D, Herman T, Zoetewei D, Ginis P, Brozgol M, Cornejo Thumm P, Decaluwe E, Ganz N, Palmerini L, Giladi N, Nieuwboer A, Hausdorff JM. Daily-Living Freezing of Gait as Quantified Using Wearables in People With Parkinson Disease: Comparison With Self-Report and Provocation Tests. Phys Ther. 2022 Dec 6;102(12):pzac129. doi: 10.1093/ptj/pzac129. PMID 36179090
- [Derived] Zoetewei D, Herman T, Brozgol M, Ginis P, Thumm PC, Ceulemans E, Decaluwe E, Palmerini L, Ferrari A, Nieuwboer A, Hausdorff JM. Protocol for the DeFOG trial: A randomized controlled trial on the effects of smartphone-based, on-demand cueing for freezing of gait in Parkinson's disease. Contemp Clin Trials Commun. 2021 Jun 29;24:100817. doi: 10.1016/j.conctc.2021.100817. eCollection 2021 Dec. PMID 34816053